CLINICAL TRIAL: NCT00630786
Title: A Phase 1b/2 Trial of AMG 655 in Combination With Panitumumab in Subjects With Metastatic Colorectal Cancer
Brief Title: Conatumumab/Panitumumab Combination Metastatic Colorectal Cancer Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060332; 2007-004722-25 (EudraCT Number)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Colon Cancer; Colorectal Cancer; Rectal Cancer; Metastatic Colorectal Cancer; Oncology
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms; Neoplasms | interventions — Panitumumab; conatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab plus conatumumab (Experimental): Participants received 10 mg/kg conatumumab and 6 mg/kg panitumumab administered on the same day by sequential intravenous (IV) infusions once every 2 weeks until progressive disease, intolerability, withdrawal, or death.
  Interventions: Drug: Panitumumab; Drug: Conatumumab

INTERVENTIONS:
Drug: Panitumumab — Administered by intravenous infusion
  Other Names: Vectibix®
Drug: Conatumumab — Administered by intravenous infusion
  Other Names: AMG 655

SUMMARY:
This is an exploratory phase 1b/2, global, multicenter, single-arm, 2-part (phase 1b and 2) study of conatumumab in combination with panitumumab in patients with Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
This is an exploratory phase 1b/2, global, multicenter, single-arm, 2-part (phase 1b and 2) study of conatumumab in combination with panitumumab in patients with Metastatic Colorectal Cancer.

The objective for Part 1 is to identify a tolerable dose of conatumumab in combination with panitumumab based on the incidence of dose-limiting toxicities in patients with Metastatic Colorectal Cancer.

The objective for Part 2 is to evaluate the objective response rate stratified by Kirsten Rat Sarcoma Virus Oncogene (KRAS) status (wild-type versus mutant) in patients with Metastatic Colorectal Cancer treated with the combination of panitumumab and conatumumab (tolerable dose identified in part 1).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the colon or rectum
* Radiographically documented disease progression per modified Response Evaluation Criteria in Solid Tumors (RECIST) during or following treatment with fluoropyrimidine, irinotecan, and/or oxaliplatin chemotherapy for Metastatic Colorectal Cancer. Progressive disease must be documented during or ≤ 6 months after the last dose of the most recent chemotherapy regimen prior to enrollment.
* At least 1 uni-dimensionally measurable lesion measuring ≥ 20 mm in one dimension per modified RECIST. Lesion must not be chosen from a previously irradiated field, unless there has been documented disease progression in that field after irradiation and prior to enrollment. All sites of disease must be evaluated.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Available archived paraffin-embedded tumor tissue from the primary tumor or metastasis for submission to the central laboratory
* Man or woman ≥ 18 years of age at the time of enrollment
* Hematologic function within the following limits:

  * Absolute neutrophil count (ANC) > 1.0 x 10^9 cells/L
  * Platelets ≥ 100 x 10^9/L
* Renal function within the following limits:

  * Creatinine < 2.0 mg/dL
* Hepatic function within the following limits:

  * Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN) (≤ 5 x ULN if liver metastases)
  * Alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases)
  * Bilirubin ≤ 2 x ULN
* Metabolic function within the following limits:

  * Amylase ≤ 2 x ULN
  * Lipase ≤ 2 x ULN
  * Magnesium ≥ lower limit of normal
* Negative pregnancy test ≤ 72 hours before enrollment (for woman of childbearing potential only)
* Must have received 1, 2, or 3 prior chemotherapy regimens for Metastatic Colorectal Cancer
* Competent to comprehend, sign, and date the independent ethics committee/institutional review board (IEC/IRB) approved written informed consent

Exclusion Criteria:

* History of other primary cancer, unless:

  * Curatively resected non-melanomatous skin cancer
  * Curatively treated cervical carcinoma in situ
  * Other primary solid tumor curatively treated with no known active disease present and no treatment administered for ≥ 5 years before enrollment
* Prior treatment with anti-epidermal growth factor receptor (EGFr) inhibitors (eg, cetuximab, erlotinib, gefitinib), unless treatment was received in the adjuvant setting ≥ 6 months before enrollment
* Use of systemic chemotherapy and radiotherapy ≤ 30 days before enrollment
* Use of prior anti-tumor therapies with a short serum half-life (less than 1 week) including prior experimental agents or approved anti-tumor small molecules ≤ 30 days before enrollment
* Use of anti-tumor therapies with a longer serum half-life (eg, bevacizumab) including prior experimental or approved protein/antibodies ≤ 42 days before enrollment
* Any investigational agent or therapy ≤ 30 days before enrollment
* Known allergy or hypersensitivity to any component of panitumumab and/or AMG 655
* History of or known presence of central nervous system (CNS) metastases
* History of interstitial lung disease (eg, pneumonitis, pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest computerized tomography (CT) scan
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment
* Active inflammatory bowel disease or other active bowel disease causing chronic diarrhea (defined as ≥ Common Terminology Criteria for Adverse Events [CTCAE] grade 2 [CTCAE version 3.0])
* Known positive test for human immunodeficiency virus (HIV) infection, hepatitis C virus, acute or chronic hepatitis B infection
* Any co-morbid disease or condition that could increase the risk of toxicity (eg, significant ascites, significant pleural effusion)
* Any uncontrolled concurrent illness (eg, infection, bleeding) or history of any medical condition that may interfere with the interpretation of the study results
* Major surgical procedure (requiring general anesthesia) ≤ 28 days or minor surgical procedure (excluding central venous catheter placement) ≤ 14 days before enrollment. Patients must have recovered from surgery related toxicities.
* Other investigational procedures are excluded
* Patient is currently pregnant or breast feeding
* Man or woman of childbearing potential who is not willing to use adequate contraceptive precautions during treatment and for 6 months (for women) or 1 month (for men) after the last investigational product administration. Adequate contraceptive precautions includes double barrier contraceptive methods (eg, diaphragm and condom) or abstinence.
* Previously enrolled into this study
* Patient unwilling or unable to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 12 January 2008 through 6 November 2008
Groups:
- Wild-type KRAS: Participants with wild-type Kirsten Rat Sarcoma Virus Oncogene (KRAS) received 10 mg/kg conatumumab and 6 mg/kg panitumumab administered on the same day by sequential intravenous (IV) infusions once every 2 weeks until progressive disease, intolerability, withdrawal, or death.
- Mutant KRAS: Participants with mutant Kirsten Rat Sarcoma Virus Oncogene (KRAS) received 10 mg/kg conatumumab and 6 mg/kg panitumumab administered on the same day by sequential intravenous (IV) infusions once every 2 weeks until progressive disease, intolerability, withdrawal, or death.
- Unknown KRAS: Participants with unknown Kirsten Rat Sarcoma Virus Oncogene (KRAS) type received 10 mg/kg conatumumab and 6 mg/kg panitumumab administered on the same day by sequential intravenous (IV) infusions once every 2 weeks until progressive disease, intolerability, withdrawal, or death.
Period: Overall Study
Arm/Group | Wild-type KRAS | Mutant KRAS | Unknown KRAS
Started | 19 (Includes 2 patients enrolled in Part 1 and 17 patients enrolled in Part 2.) | 25 (Includes 3 patients enrolled in Part 1 and 22 patients enrolled in Part 2.) | 9 (All patients were enrolled in Part 2.)
Received Study Medication | 19 | 25 | 8
Completed | 18 (Completed study defined as participant death) | 23 (Completed study defined as participant death) | 7 (Completed study defined as participant death)
Not Completed | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wild-type KRAS | Mutant KRAS | Unknown KRAS | Total
Number analyzed (Participants) | 19 | 25 | 8 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.53 (12.53) | 64.32 (12.35) | 58.63 (13.65) | 62.42 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 3 | 27
  Male | 6 | 14 | 5 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  White or Caucasian | 16 | 24 | 7 | 47
  Black or African American | 3 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose-limiting Toxicities
Description: A dose-limiting toxicity (DLT) was defined as any grade 3 or 4 conatumumab-related or combination (panitumumab and conatumumab)-related adverse event, or grade 3 or 4 laboratory abnormality that occurred during the first 4 weeks (28 days) of treatment with panitumumab and conatumumab. Anemia and lymphopenia were not considered DLTs.
  Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was used to grade all adverse events and toxicities.
Time Frame: 4 weeks
Population: DLT-evaluable patients were those who received ≥ 2 doses of panitumumab and conatumumab as scheduled (ie, weeks 1 and 3) and completed 4 weeks (28 days) of treatment, or had a DLT within the first 4 weeks (28 days) of treatment.
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus Conatumumab
Number analyzed (Participants) | 5
participants | 0

2. Primary Outcome: Number of Participants With an Objective Response
Description: An overall objective response of either a confirmed complete response or partial response, where the overall objective response was equivalent to the best overall response recorded for each participant from enrollment until disease progression or recurrence. Tumor response was assessed by the investigator according to the modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. Responses were confirmed no less than 4 weeks after the criteria for response were first met. Complete response defined as the disappearance of all target and non-target lesions and no new lesions. Partial response defined as either the disappearance of all target lesions with the persistence of one or more non-target lesion(s), or, at least a 30% decrease in the sum of the longest diameter (SLD) of target lesions, taking as reference the Baseline SLD and the disappearance of all or the persistence of 1 or more non-target lesions.
Time Frame: Participants were evaluated for tumor response until radiographic disease progression or until the participant began another anticancer treatment (up to a maximum of 55.6 weeks).
Population: Subset of the Safety Analysis Set, composed of all enrolled participants who received at least one dose of study drug who had known Kirsten Rat Sarcoma Virus Oncogene (KRAS) status and Baseline measurable disease.
Measure: Number; unit: participants
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 18 | 25
participants | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier estimate of the median time from enrollment to death from any cause or disease progression. Progressive disease is defined as at least a 20% increase in the sum of the longest diameters (SLD) of target lesions, taking as reference the nadir SLD recorded since the treatment started, or the appearance of one or more new lesions, or the unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 2
Population: Subset of the Safety Analysis Set, composed of all enrolled participants who received at least one dose of study drug who had known Kirsten Rat Sarcoma Virus Oncogene (KRAS) status.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 19 | 25
weeks | 10.0 [7.0 to 23.0] | 7.1 [6.7 to 8.0]

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimate of time from enrollment to death from any cause
Time Frame: as for outcome 2
Population: Subset of the Safety Analysis Set, composed of all enrolled participants who received at least one dose of study drug, who had known Kirsten Rat Sarcoma Virus Oncogene (KRAS) status.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 19 | 25
months | 7.3 [3.2 to 15.0] | 4.4 [3.4 to 8.5]

5. Secondary Outcome: Number of Participants With Disease Control
Description: Disease control defined as participants with an overall objective response of complete response (CR), partial response (PR), or stable disease during the treatment period, assessed by the investigator according to the modified Response Evaluation Criteria in Solid Tumors (RECIST). Responses were confirmed no less than 4 weeks after the criteria for response were first met. CR defined as the disappearance of all target and non-target lesions and no new lesions. PR defined as either the disappearance of all target lesions with the persistence of one or more non-target lesion(s), or, at least a 30% decrease in the sum of the longest diameter (SLD) of target lesions, taking as reference the Baseline SLD and the disappearance of all or the persistence of 1 or more non-target lesions. Stable disease defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the nadir LD since the treatment started.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 19 | 25
participants | 8 | 4

6. Secondary Outcome: Time to Response
Description: The interval in days from the first dose of study therapy to the date of first confirmed objective response. Calculated only for participants with an objective response.
Time Frame: as for outcome 2
Population: Patients with an overall objective response
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duation of Response
Description: The interval in days from the first confirmed objective response to disease progression per the modified RECIST criteria or death. Calculated only for participants with an objective response.
Time Frame: as for outcome 2
Population: Patients with an overall objective response
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Anti-therapeutic Antibodies
Description: Number of participants with human anti-panitumumab antibodies (HAPA) or anti-conatumumab antibodies measured by immunoassay.
Time Frame: Antibody samples were collected at weeks 1, 7, and 23 and every 6 months thereafter during treatment, and at the safety follow-up and follow-up visits. The mean follow-up time was 35.7 weeks.
Population: Safety analysis set, including all randomized patients who received at least 1 dose of investigational product. N indicates the number of patients with immunoassay results at the specified time points.
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus Conatumumab
Number analyzed (Participants) | 52
participants
  Anti-panitumumab Antibody at Baseline (N=51) | 0
  Anti-panitumumab Antibody Post-baseline (N=37) | 2
  Anti-conatumumab Antibody at Baseline (N=50) | 1
  Anti-conatumumab Antibody Post-baseline (N=37) | 0

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment, and includes any such occurrence (eg, sign, symptom, or diagnosis) or worsening of a pre-existing medical condition from the time that a participant has signed informed consent to the time of initiation of investigational product. The severity of AEs was graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, according to the following:
  1. = Mild: Aware of sign or symptom, but easily tolerated
  2. = Moderate: Discomfort enough to cause interference with usual activity;
  3. = Severe: Incapacitating with inability to work or do usual activity;
  4. = Life-threatening: an event in which the patient was, in the view of the investigator, at risk of death at the time of the event;
  5. = Fatal.
Time Frame: From first dose of investigational drug until 30 days after the last dose, up to a maximum of 50 weeks.
Population: Safety Analysis Set, including all randomized patients who received at least one dose of investigational drug.
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus Conatumumab
Number analyzed (Participants) | 52
participants
  Any adverse event | 51
  Grade 3 adverse event | 16
  Grade 4 adverse event | 4
  Grade 5 adverse event | 6

10. Secondary Outcome: Number of Participants With Post-baseline Laboratory Values Grade 3 or Higher
Description: Laboratory values were assessed using the National Cancer Institute (NCI) Common Toxicity Criteria (version 3.0) according to the following: 1 = Mild; 2 = Moderate; 3 = Severe; 4 = Life-threatening; 5 = Fatal.
Time Frame: From first dose of investigational drug until 30 days after the last dose, up to a maximum of 50 weeks.
Population: Safety Analysis Set, including all randomized patients who received at least one dose of investigational drug.
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus Conatumumab
Number analyzed (Participants) | 52
participants
  Alanine Amino Transferase increase | 4
  Alkaline Phosphatase increase | 9
  Amylase increase | 2
  Aspartate Amino Transferase increase | 5
  Bicarbonate decrease | 1
  Calcium increase | 1
  Calcium decrease | 3
  Glucose increase | 1
  Lipase increase | 2
  Magnesium decrease | 4
  Magnesium increase | 1
  Phosphorus decrease | 1
  Sodium decrease | 1
  Total Bilirubin increase | 6
  Absolute Neutrophil Count decrease | 7
  Hemoglobin decrease | 4
  Lymphocytes decrease | 7

ADVERSE EVENTS:
Time Frame: From first dose of investigational drug until 30 days after the last dose, up to a maximum of 50 weeks.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Panitumumab + AMG 655
Serious Adverse Events (participants affected / at risk) | 26/52
Other Adverse Events (participants affected / at risk) | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + AMG 655 (N=52)
Atrial fibrillation (Cardiac disorders) | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pneumoperitoneum (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 2
General physical health deterioration (General disorders) | 4
Performance status decreased (General disorders) | 1
Pyrexia (General disorders) | 4
Bile duct obstruction (Hepatobiliary disorders) | 1
Biliary dilatation (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Abdominal wall abscess (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab + AMG 655 (N=52)
Anaemia (Blood and lymphatic system disorders) | 3
Growth of eyelashes (Eye disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 9
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 16
Oral pain (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 17
Asthenia (General disorders) | 7
Chills (General disorders) | 7
Fatigue (General disorders) | 20
Mucosal inflammation (General disorders) | 10
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 5
Pyrexia (General disorders) | 9
Folliculitis (Infections and infestations) | 5
Paronychia (Infections and infestations) | 6
Procedural pain (Injury, poisoning and procedural complications) | 3
Weight decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dysgeusia (Nervous system disorders) | 3
Neuralgia (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Acne (Skin and subcutaneous tissue disorders) | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 10
Erythema (Skin and subcutaneous tissue disorders) | 12
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 28
Scab (Skin and subcutaneous tissue disorders) | 7
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.